CLINICAL TRIAL: NCT01509352
Title: Prospective Randomized Trial Evaluating the Utility of Esophageal Stitches During Laparoscopic Fundoplication.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10 01-003
Record Dates: First submitted 2011-12-14; First posted 2012-01-13 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Reflux
Keywords: fundoplication; gastric reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with esophageal stitches (Active Comparator): fundoplication with crural stitches
  Interventions: Procedure: esophageal stitches during fundoplication
- without esophageal stitches (Experimental): fundoplication without crural stitches.
  Interventions: Procedure: no esophageal stitches placed during fundoplication

INTERVENTIONS:
Procedure: esophageal stitches during fundoplication — placement of esophageal stitches with fundoplication
  Other Names: crural stitches.
  Arms: with esophageal stitches
Procedure: no esophageal stitches placed during fundoplication — no esophageal stitches are placed during the fundoplication procedure
  Other Names: crural stitches
  Arms: without esophageal stitches

SUMMARY:
This is a prospective trial of the utility of esophageal stitches during fundoplication.

The hypothesis is that recurrence rate may be different with or without the esophageal stitches.

DETAILED DESCRIPTION:
This will be a single center, prospective randomized clinical trial involving patients who require an operation for gastroesophageal reflux disease. This is intended to be a definitive study. All patients will receive the standard operation for reflux: laparoscopic fundoplication. The dissection will be performed by leaving the phrenoesophageal membrane intact in all patients.

One group will undergo laparoscopic fundoplication with 4 esophageal-crural sutures while the other group will not have these placed. The operation, post-operative care, and follow-up plan will otherwise not differ between groups.

ELIGIBILITY:
Inclusion Criteria:

Patients less than 7 years of age requiring fundoplication for gastroesophageal reflux disease who are considered good laparoscopic candidates by the staff surgeon will be considered candidates.

Exclusion Criteria:

1. Hiatal hernia demonstrated on preoperative contrast study, computed tomography, endoscopy, or intraoperative findings.
2. Prior esophageal operation (e.g. esophageal atresia repair, esophageal myotomy)
3. Prior operation for congenital diaphragmatic hernia
4. Patients not considered laparoscopic candidates by the staff surgeon or anesthesiologist (e.g. carbon dioxide retaining lung disease, congenital heart disease, or complex previous abdominal operations)

Ages: 1 Day to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2010-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
hiatal herniation | 4 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No